CLINICAL TRIAL: NCT06598904
Title: The Effect of Aromatherapy on Anxiety and Pain for First Dental Visit Patients: a Randomized Controlled Clinical Trial
Brief Title: The Effect of Aromatherapy for First Dental Visit Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, He Cai, Post Doctor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WCHS-CRSE-2024-128-R1-P
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; aromatherapy; first dental visit

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: single-note lavender essential oil (Experimental): Aroma diffuser with single-note lavender essential oil.
  Interventions: Other: Aroma diffuser with single-note lavender essential oil
- Group 2: single-note orange essential oil (Experimental): Aroma diffuser with single-note orange essential oil
  Interventions: Other: Aroma diffuser with single-note orange essential oil
- Group 3: deionized water (Placebo Comparator): Aroma diffuser with deionized water.
  Interventions: Other: Aroma diffuser with deionized water

INTERVENTIONS:
Other: Aroma diffuser with single-note lavender essential oil — In a space of 3*4*2.6 cubic meters, positioned 10 cm away from the patient, add 4-6 drops (each drop being 0.05 ml) of 100% concentration single-note lavender essential oil into the aroma diffuser reservoir containing 120 ml of water.
  Arms: Group 1: single-note lavender essential oil
Other: Aroma diffuser with single-note orange essential oil — In a space of 3*4*2.6 cubic meters, positioned 10 cm away from the patient, add 4-6 drops (each drop being 0.05 ml) of 100% concentration single-note orange essential oil into the aroma diffuser reservoir containing 120 ml of water.
  Arms: Group 2: single-note orange essential oil
Other: Aroma diffuser with deionized water — In a space of 3*4*2.6 cubic meters, positioned 10 cm away from the patient, add 4-6 drops (each drop being 0.05 ml) of water into the aroma diffuser reservoir containing 120 ml of deionized water.
  Arms: Group 3: deionized water

SUMMARY:
First dental visit experience is strongly correlated with dental anxiety, the aim of this protocol is to explore the efficacy of olfactory aromatherapy for the reduce of dental anxiety and pain in first-visit patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who never visited dental clinics before;
* Patients who need dental treatment, such as resin filling, root canal treatment, periodontal initial treatment, tooth extraction, etc;
* Patients and their guardians who are able to understand the purpose of the study and volunteer to take part in the study;
* Patients who are intellectually sufficient to complete the anxiety scale;
* Be able to complete all assessments and follow-up during the study.

Exclusion Criteria:

* Patients who are allergic to the ingredients of the essential oils used in the experiment or to the materials used in the dental treatment;
* Patients who underwent only an oral examination;
* Patients with severe heart disease, hypertension, respiratory disease, or other systemic conditions that were not eligible for trial participation;
* Pregnant or lactating women;
* People with depressive symptoms, anxiety disorders or other mental illnesses that affect their mood state;
* People who are using sedative or analgesic drugs;
* Recent or current users of essential oils;
* Any circumstances considered by the investigator to be inappropriate for participation in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety scale 1 - Modified Dental Anxiety Scale (MDAS) | 5 minutes before operation/during operation (immediately after the most painful procedure)/immediately after operation.
  The Modified Dental Anxiety Scale (MDAS) consists of 4 questions each with a 5 category rating scale, ranging from 'not anxious' to 'extremely anxious', hence, the total score varies from 4 to 20, with higher obtained scores describing more elevated levels of dental anxiety. MDAS is recorded before, during and after operation.
Pain scale - Visual Analog Scale (VAS) | 5 minutes before operation/during operation (immediately after the most painful procedure)/immediately after operation.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." VAS is recorded before, during and after operation.

SECONDARY OUTCOMES:
Anxiety scale 2 - State-Trait Anxiety Inventory for State Anxiety (STAI-S) | 5 minutes before operation/ immediately after operation.
  The STAI-S evaluates the subjective feelings of tension, worry, nervousness, apprehension, and autonomic nervous system activation. This self-completed inventory consisted of 20 items on a four-point Likert scale running from one (i.e., not at all) to four (i.e., very much). Hence, the total score varies from 20 to 80, with higher obtained scores describing more elevated levels of anxiety. STAI-S is recorded before and after operation.
Vital sign 1 - systolic blood pressure (SBP) | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation.
  Systolic blood pressure (SBP) is measured using a manual sphygmomanometer, before, during and after operation.
Vital sign 2 - diastolic blood pressure (DBP) | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation.
  Diastolic blood pressure (DBP) is measured using a manual sphygmomanometer, before, during and after operation.
Vital sign 3 - heart rate (HR） | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation.
  Heart rate (HR) is measured as pulse rate using an oximeter, before, during and after operation.
Vital sign 4 - oxygen saturation (SpO2） | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation.
  Oxygen saturation (SpO2）is measured using an oximeter, before, during and after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology SIchuan University, Chengdu, Sichuan, China